CLINICAL TRIAL: NCT01677663
Title: Neuropsychopathological Study of Autism: From Clinical, Neurocognitive, to Genetic Studies and Animal Models
Brief Title: Neuropsychopathological Study of Autism
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Taiwan University (Other)
Responsible Party: Principal Investigator, National Taiwan University Hospital, Susan Shur-Fen Gau, National Taiwan University Hospital
Other Study IDs: 201103003RB
Record Dates: First submitted 2012-08-30; First posted 2012-09-03 (Estimated); Last update posted 2012-09-03 (Estimated); Status verified 2012-08

CONDITIONS: Autism
Keywords: autism; clinical phenotypes; neuropsychology; imaging endophenotypes; family-based cohort; knoutout mice
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Observational Model: Family Based
Biospecimen Retention: Samples With DNA — The subjects will receive blood withdrawal. The blood sample will be used for establishing lymphoblastoid cell lines, which will be used for molecular genetic experiments.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Autism or autism spectrum disorder (ASD) is a relatively common (0.3% in Taiwan), multi-factorial, genetically and clinically heterogeneous, childhood-onset neurodevelopmental disorder. Due to its high heritability and severe long-term impairment without available laboratory diagnosis, effective prevention or treatment, this disastrous disease has been prioritized for molecular genetic studies. Recent CNVs investigation to identify rare variants and GWA study with endophenotype approaches are promising strategies to identify common genetic variants. In addition to intermediate phenotypes such as head circumstance, speech delay, social impairments and stereotyped behaviors, evidence has demonstrated that neuropsychology and neuroimages may be useful endophenotypes for autism. Dlgap2, Fbxo25, and Arhgef10 knoutout mice generated from our previous CNV results will be characterized.

DETAILED DESCRIPTION:
The specific aims of the study aree:

1. To collect complete environmental, developmental, clinical, neuropsychological, and genetic data of 350 probands with autism (800 in total, 450 from [96HD008]) and their families;
2. To re-sequence promoter region, all the exons, and the 3'UTR region of the DLGAP2, CLN8, ARHGEF10, FBXO25, and GABRB3 genes (one gene per year);
3. To conduct fine-mapping and replication studies for selected candidate genes from GWA study[96HD008];
4. To validate social impairment and speech delay as intermediate phenotypes and the executive functions as effective cognitive endophenotypes by first demonstrating the differences in these measures among probands, their unaffected siblings and neurotypicals, followed by different genetic risks (e.g., neurexin, neuroligin, CNTNAP2, SHANK3, MET, PTEN, WNT2, FOXP2, DLGAP2, CLN8, ARHGEF10, FBXO25, and GABRB3);
5. To validate the structural and functional connectivity as effective imaging endophenotypes by demonstrating the differences between probands with autism, their siblings, and matched neurotypicals; and
6. To characterize the phenotypes of and to explore the possible function of other autism-related genes found by using GWAS, and to explore the possible drug targets for the treatment for Dlgap2, Fbxo25, and Arhgef10 mutant mice.

The investigators will recruit 350 probands with clinical diagnosis of autism confirmed by the ADI-R and ADOS, and their families. The probands and their siblings will also be assessed for other psychiatric disorders (K-SADS-E); autistic symptom dimensions (SRS, SCQ, CAST, ABC), other behavioral symptoms (CBCL, SNAP-IV), and perinatal/environmental risk factors. The direct tests include intelligence (CPM/SPM, WISC-III, WPPSI-R) and neuropsychological tests (CPT, WCST, CANTAB). The parents will be assessed for DSM-IV psychiatric disorders (ASRI-4) and autistic features (AQ, SRS). The investigators will collect blood samples from all the subjects. Probands with previous CNVs findings (n = 20) and high-functioning autism (n=30) will receive the MRI assessments (Diffusion Spectrum Imaging, resting-state fMRI) as compared to 50 age-, sex-, and handedness-matched neurotypicals.

The investigators will (1) characterize the behavioral, structural, electrophysiological and biochemical phenotypes of Dlgap2, and Arhgef10 mice at 4 weeks, 8 weeks, 12 weeks and 16 weeks of ages; (2) explore the possible function of other autism-related genes found by GWAS analysis; and (3) explore the possible drug targets for the treatment of autism from KO mice. While the potential target is recognized, existing compounds of this target can be tested.

The investigators anticipate to establishing a representative cohort of 800 patients with autism and their families from this study and [96HD008] with comprehensive clinical and genetic data. This well-characterized cohort will contribute to validation of intermediate phenotypes and cognitive and imaging endophenotypes for autism in this study, and will be used to search for rare variants by CNVs analysis and common variants by GWAS analysis in future study, and will pave the way to have 2-3 lines of well-characterized transgenic animal models of autism (e.g., Dlgap2). In addition, a wealth of data from this cohort will benefit to current and future investigation on autism and will be the basis for future international collaboration. The investigators also anticipated to publication of 20 SCI papers (4 per year) and presentation of our work in peer-reviewed scientific conferences by more than 40 posters or oral communications.

ELIGIBILITY:
Inclusion Criteria:

* subjects have a clinical diagnosis of autistic disorder or Asperger disorder defined by the DSM-IV and ICD-10;
* their ages range from 3 to 25 when we conduct the study;
* subjects have at least one biological parent;
* both parents of the subjects are Han Chinese;
* subjects and their biological parents (and siblings if any) consent to participate in this study.

Exclusion Criteria:

* if they currently meet criteria or have a history of DSM-IV Schizophrenia, Schizoaffective Disorder, or Organic Psychosis.

Ages: 3 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The sample will consist of 350 probands with ASD, aged 3-25.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2011-08; Study Completion 2016-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Shur-Fen Gau, MD, PhD, Principal Investigator — National Taiwan University Hospital & College of Medicine
Locations (1):
- National Taiwan Univeristy Hospital, Taipei, Taiwan